CLINICAL TRIAL: NCT00469950
Title: Effect of Exercise Training After Percutaneous Coronary Intervention
Brief Title: The Effect of Training on Endothelial Function, Progression of Disease,Inflammation, Heart Rate Variability and Mental Health After Percutaneous Coronary Intervention
Acronym: EFECTOR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3.2005.1437
Record Dates: First submitted 2007-05-04; First posted 2007-05-07 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2009-02

CONDITIONS: Coronary Artery Disease
Keywords: PCI; stent; training; endothelial function; restenosis; late luminal loss; heart rate variability; oxygen uptake capacity; inflammatory markers
MeSH Terms: conditions — Coronary Artery Disease | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: exercise training — Exercise training in groups

SUMMARY:
The Efector study is an open, randomized and controlled trial assessing the effect of regular exercise training on endothelial function, inflammatory markers, progression of disease, heart rate variability and mental health in patients who have been successfully treated with percutaneous coronary intervention and stent implantation for angina pectoris.

DETAILED DESCRIPTION:
Pas er randomized to a 6 months training group or none training. At baseline and at 6 months patients are examined with blood tests to measure serum concentrations of inflammatory markers, a test for endothelial function, heart rate variability and a coronary angiogram. Further patients are asked to answer questionnaires concerning mental health (SF36, HADS).

ELIGIBILITY:
Inclusion Criteria:

* Successful PCI with stent implantation,
* Able to participate in the training program,
* No planned further revascularisation

Exclusion Criteria:

* CAGB,
* Inflammatory diseases other than CAD,
* Heart failure,
* Severe kidney failure,
* Inability to participate in the training program

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
flow mediated dilation, serum concentrations of biomarkers, restenosis-rate/ late luminal loss, heart rate variability in SDNN | 6 months

SECONDARY OUTCOMES:
Oxygen uptake capacity (mg/kg/min), Sf36 scores | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Munk, MD, Principal Investigator — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Stavanger, Rogaland, Norway

REFERENCES:
- [Derived] Munk PS, Breland UM, Aukrust P, Ueland T, Kvaloy JT, Larsen AI. High intensity interval training reduces systemic inflammation in post-PCI patients. Eur J Cardiovasc Prev Rehabil. 2011 Dec;18(6):850-7. doi: 10.1177/1741826710397600. Epub 2011 Feb 18. PMID 21450602
- [Derived] Munk PS, Staal EM, Butt N, Isaksen K, Larsen AI. High-intensity interval training may reduce in-stent restenosis following percutaneous coronary intervention with stent implantation A randomized controlled trial evaluating the relationship to endothelial function and inflammation. Am Heart J. 2009 Nov;158(5):734-41. doi: 10.1016/j.ahj.2009.08.021. PMID 19853690